CLINICAL TRIAL: NCT04228640
Title: A Multicentre, Randomized, Double Blind, Parallel Design, Placebo Controlled Study to Evaluate the Efficacy and Safety of Uthever (NMN), an Orally Administered Supplementation in Middle Aged and Older Adults.
Brief Title: Evaluate the Efficacy and Safety of Uthever NMN(Nicotinamide Mononucleotide, a Form of Vitamin B3)
Acronym: NMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EffePharm LTD (Industry)
Collaborators: ProRelix Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFFE-CT-01
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Aging
Keywords: Anti- Aging; Workout Enhancer

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator
Masking Description: Randomized, Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): Ingredient: NMN Dosage form: Capsule, 150 mg/capsule Frequency: 2 capsules per day Duration: 60 days
  Interventions: Other: NMN
- Placebo (Placebo Comparator): Ingredient: Starch powder Dosage form: Capsule, 150 mg/capsule Frequency: 2 capsules per day Duration: 60 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: NMN — Investigational Product
  Arms: Investigational Product
Other: Placebo — Starch Powder
  Arms: Placebo

SUMMARY:
This will be a multi-center, two arm study in 66 healthy adults. Subjects will complete a screening visit (V1, Day -7) to determine eligibility for the study based on Inclusion & Exclusion Criteria, patient history and safety measures. Eligibility confirmation will be done on visit 2 (Day 1). Patients successfully completing screen will be assigned to either of the two treatments. Subjects will receive the treatment for at-home use and will also be given diaries for recording information of medication, and adverse events. At 2 different intervals i.e. Day 30 and Day 60 (V3, V4) subjects will return to the clinic to review and collect patient diaries, safety data and medication reconciliation. Efficacy and safety assessments will be done at baseline, Day 30 and Day 60 .

DETAILED DESCRIPTION:
Sixty-six healthy male or female middle-aged or older subjects will be assigned in 1:1 ratio to treatment with the test product, NMN or Placebo in this double-blind, randomized, placebo-controlled study. All 66 enrolled subjects will be instructed to take two capsules of either NMN or Placebo once a day after breakfast for 60 days daily. Subjects will be required to use diaries to document the date and time of study treatments including any missed doses and the occurrence of any adverse events.

The duration of each subject's participation in the study will be of 60 days.

Scheduled study visits will include:

* Visit 1 (Screening, Day -4)
* Visit 2 (Baseline/Randomization visit, Day 1)
* Visit 3 (Day 30).
* Visit 4 (End of study, Day 60) A window (± 2 days) will be considered acceptable for each scheduled visit following the baseline visit.

During Visit 1 (Screening), informed consent will be obtained before any study procedures take place. After subject has been consented, medical history will then be documented, including the concomitant medications (if any). Physical examination and ECG will be carried out for all subjects. Subjects' vital signs will be recorded along with pulse pressure (PP).Their laboratory investigations like Hematology, Clinical chemistry and Urinalysis will be done. They shall undergo the screening procedure by inclusion and exclusion criteria. Subject's demography data will be collected. They will be given instructions for the next visit.

At Visit 2 (Day 1, Baseline visit), eligibility confirmation will be done, and each enrolled subject will be randomly assigned in double-blind fashion, in 1:1 ratio to the test product or the Placebo. Blinded investigational product will be dispensed to subjects who meet all the inclusion and none of the exclusion criteria. Subjects will be instructed to take two capsules of the either placebo or NMN once a day with ambient temperature water after breakfast. They shall be recording the dosing details in subject diaries. The first dose of Investigational Product will be taken by the subject at home. Subjects will be evaluated through SF-36 questionnaire for their health. They will be required to answer few questions pertaining to their health. (PI, CRC or site staff will fill SF-36 questionnaire in visit 2, 3 and 4 by asking the subject). All the baseline assessments for efficacy will be performed.

At visit 3 (Day 30) and visit 4 (Day 60), subjects will return to the clinic to review and collect subjects' diaries, safety data, and medication reconciliation. Efficacy and safety assessments will be done at both the visits.

Subjects will be asked to bring their subject diaries and used/unused Investigational Products every time they visit the site. Enough quantity of Investigational Product will be dispensed every visit. Subjects' vital signs will be recorded along with pulse pressure (PP) at all visits. Adverse event assessment and concomitant assessment will be done at each visit along with compliance with drug applications.

ELIGIBILITY:
Inclusion Criteria:

1. Male/females of 40 to 65 years of age
2. Body Mass Index (BMI) between 18.5 and 35 kg/m2
3. Able to provide written Informed Consent
4. Able to follow verbal and written study directions
5. Must not be taking or be willing to take any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.
6. Able to maintain consistent diet and lifestyle habits throughout the study
7. Male and female subjects must be willing to agree to use effective contraceptive methods while on treatment and for 3 months after the completion of study
8. Willing to consume assigned dietary supplements for 2 months

Exclusion Criteria:

1. Participants on current use of prescription or over-the-counter nicotinic acid
2. Use of statin drugs
3. Having used any tobacco product or used a recreational drug in the past 6 months
4. Having abnormal screening laboratory test values or other lab test result(s) that would preclude study participation in the judgment of the investigator
5. Documented presence of atherosclerotic disease and/or cardiopulmonary disease
6. History of drug or alcohol abuse
7. History of unstable depression or mental illness within the last 6 months for which the investigator believes could impact the participant's ability to comply with study requirements
8. Unwilling to discontinue use of conventional multivitamin/mineral or other supplements at least two weeks prior to the study start
9. Participating in or planning to begin a weight loss diet during the study period
10. Chronic use of over-the-counter medication which would interfere with study endpoints
11. Lifestyle or schedule incompatible with the study protocol
12. Known hypersensitivity to the drug components used during the study
13. Women with positive result for urinary beta human chorionic gonadotropin or gestation period or breastfeeding
14. Other diseases or medications, according to the investigator, that would interfere directly in the results of the study or jeopardize the health of the participant.
15. Currently, or within the past 30 days, enrolled in a different clinical investigation
16. Inability to provide a venous blood sample
17. Unable or unwilling to provide written informed consent for participation in study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Blood cellular NAD+ concentration in serum | Day 2
  Evaluation of Blood cellular NAD+ concentration in serum inter group comparison from baseline to the end of study
Blood cellular NAD+ concentration in serum | Day 30
  Evaluation of Blood cellular NAD+ concentration in serum inter group comparison from baseline to the end of study
Blood cellular NAD+ concentration in serum | Day 60
  Evaluation of Blood cellular NAD+ concentration in serum inter group comparison from baseline to the end of study
Blood cellular NADH concentration in serum | Day 2
  Evaluation of Blood cellular NADH concentration in serum inter group comparison from baseline to the end of study
Blood cellular NADH concentration in serum | Day 30
  Evaluation of Blood cellular NADH concentration in serum inter group comparison from baseline to the end of study
Blood cellular NADH concentration in serum | Day 60
  Evaluation of Blood cellular NADH concentration in serum inter group comparison from baseline to the end of study
Six minutes walking endurance test | Day 2
  Evaluation of Six minutes walking endurance test inter group comparison from baseline to the end of study
Six minutes walking endurance test | Day 30
  Evaluation of Six minutes walking endurance test inter group comparison from baseline to the end of study
Six minutes walking endurance test | Day 60
  Evaluation of Six minutes walking endurance test inter group comparison from baseline to the end of study
Systolic | Day 2
  Evaluation of Systolic blood pressure inter group comparison from baseline to the end of study
Systolic | Day 30
  Evaluation of Systolic blood pressure inter group comparison from baseline to the end of study
Systolic | Day 60
  Evaluation of Systolic blood pressure inter group comparison from baseline to the end of study
Diastolic blood pressure | Day 2
  Evaluation of diastolic blood pressure inter group comparison from baseline to the end of study
Diastolic blood pressure | Day 30
  Evaluation of diastolic blood pressure inter group comparison from baseline to the end of study
Diastolic blood pressure | Day 60
  Evaluation of diastolic blood pressure inter group comparison from baseline to the end of study
Pulse pressure | Day 2
  Evaluation of Pulse Pressure inter group comparison from baseline to the end of study
Pulse pressure | Day 30
  Evaluation of Pulse Pressure inter group comparison from baseline to the end of study
Pulse pressure | Day 60
  Evaluation of Pulse Pressure inter group comparison from baseline to the end of study
SF-36 questionnaire | Day 2
  Evaluation of SF-36 questionnaire inter group comparison from baseline to the end of study
SF-36 questionnaire | Day 30
  Evaluation of SF-36 questionnaire inter group comparison from baseline to the end of study
SF-36 questionnaire | Day 60
  Evaluation of SF-36 questionnaire inter group comparison from baseline to the end of study

SECONDARY OUTCOMES:
Adverse events | Day 2
  Evaluation of Adverse events
Adverse events | Day 30
  Evaluation of Adverse events
Adverse events | Day 60
  Evaluation of Adverse events
Laboratory parameter (blood chemistry) | Day 1
  Evaluation of Laboratory parameter (blood chemistry) changes from baseline to end of the study
Laboratory parameter (blood chemistry) | Day 30
  Evaluation of Laboratory parameter (blood chemistry) changes from baseline to end of the study
Laboratory parameter (blood chemistry) | Day 60
  Evaluation of Laboratory parameter (blood chemistry) changes from baseline to end of the study
Laboratory parameter (lipid profile) | Day 1
  Evaluation of Laboratory parameter (lipid profile) changes from baseline to end of the study
Laboratory parameter (lipid profile) | Day 30
  Evaluation of Laboratory parameter (blood chemistry, lipid profile, LFT and RFT) changes from baseline to end of the study
Laboratory parameter (lipid profile) | Day 60
  Evaluation of Laboratory parameter (lipid profile) changes from baseline to end of the study
Laboratory parameter (LFT ) | Day 1
  Evaluation of Laboratory parameter (LFT ) changes from baseline to end of the study
Laboratory parameter (LFT) | Day 30
  Evaluation of Laboratory parameter (LFT ) changes from baseline to end of the study
Laboratory parameter (LFT) | Day 60
  Evaluation of Laboratory parameter (LFT ) changes from baseline to end of the study
Laboratory parameter (RFT) | Day 1
  Evaluation of Laboratory parameter (RFT) changes from baseline to end of the study
Laboratory parameter (RFT) | Day 30
  Evaluation of Laboratory parameter (RFT) changes from baseline to end of the study
Laboratory parameter (RFT) | Day 60
  Evaluation of Laboratory parameter (RFT) changes from baseline to end of the study
Drop out due to adverse events | Day 2
  Number of participants that dropout due to adverse events including lab values
Drop out due to adverse events | Day 30
  Number of participants that dropout due to adverse events including lab values
Drop out due to adverse events | Day 60
  Number of participants that dropout due to adverse events including lab values

OTHER OUTCOMES:
BMI | Day 1
  Monitoring of BMI inter group comparison from baseline to the end of study
BMI | Day 2
  Monitoring of BMI inter group comparison from baseline to the end of study
BMI | Day 30
  Monitoring of BMI inter group comparison from baseline to the end of study
BMI | Day 60
  Monitoring of BMI inter group comparison from baseline to the end of study
HOMA | Day 2
  Monitoring of HOMA inter group comparison from baseline to the end of study
HOMA | Day 60
  Monitoring of HOMA inter group comparison from baseline to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Avhad, Principal Investigator — Swasthiye Clinic and Research Center
Locations (2):
- India (2):
  - Dr Kamalakar Gajarae, Pune, Maharashtra
  - Swasthiye Clinic and Research Center, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang H. A Multicentre, Randomised, Double Blind, Parallel Design, Placebo Controlled Study to Evaluate the Efficacy and Safety of Uthever (NMN Supplement), an Orally Administered Supplementation in Middle Aged and Older Adults. Front Aging. 2022 May 5;3:851698. doi: 10.3389/fragi.2022.851698. eCollection 2022. PMID 35821806